CLINICAL TRIAL: NCT04878133
Title: OCT Guided vs COmplete Pci in patieNts With sT Segment Elevation myocArdial infarCtion and mulTivessel Disease
Acronym: OCT-CONTACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Cardiologist, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCT - 001621
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Patients with STEMI who underwent successful culprit-lesion PCI will be enrolled after the index PCI. Eligible patients will be required to have residual multivessel disease, defined as at least one stenosis >
  50 %. Patients will be randomized in a 1:1 fashion to OCT guided PCI of non-culprit lesions (Group A) vs complete PCI. (Group B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exsperimental Arm (Experimental)
  Interventions: Diagnostic Test: OCT - optical coherence tomography
- Control Arm (No Intervention)

INTERVENTIONS:
Diagnostic Test: OCT - optical coherence tomography — The principle by which OCT works is similar to ultrasound, although light waves close to infrared are used instead of ultrasounds.
  In practice, the light waves, emitted into the vessel through a special catheter positioned in the coronary artery, meet the surrounding structures and are partly absorbed and partly reflected by them. The reflected waves are picked up by a sensor positioned on the catheter and analyzed through software that produces images visible live on a special console.
  Arms: Exsperimental Arm

SUMMARY:
STEMI patients with multivessel disease will be randomized to complete PCI versus PCI driven by high risk criteria of plaques evaluated with OCT

DETAILED DESCRIPTION:
In patients with ST segment elevation myocardial infarction (STEMI), percutaneous coronary intervention (PCI) of the culprit lesion significally reduces the risk of cardiovascular death. How to manage in this setting non-culprit lesion in patients with multivessel disease still remain a matter of debate. Recently, the COMPLETE trial showed that complete PCI of every coronary stenosis > 70% (or 50-69% lesions with FFR < 0.8) reduces risk of myocardial infarction (MI) and unstable angina (UA) at 3 years compared with culprit-lesion PCI [1]. Whether this findings are related to revascularization of every obstructive lesions rather than lesions with vulnerable-plaque characteristics, still remain unclear.

In high risk patients such as STEMI patients, physiopathology of coronary plaque deeply differs from stable angina, mainly due to peculiar features of plaque. STEMI lesions, when evaluated at autopsy or at intracoronary imaging, showed a pro-thrombotic pattern, with high prevalence of thin cap fibro-atheroma, plaque rupture or thrombus, and a larger amount of lipids and macrophage [2-6]. In this setting, angiography, even when combined with fractional flow reserve evaluation (which can describe more accurately the functional impact of the plaque), has intrinsic limitations because of lack of information about plaque characteristics [7,8].

Optical coherence tomography (OCT) is the latest development in intravascular coronary imaging. Similarly to intravascular ultrasound (IVUS), OCT provides cross-sectional images of the vessel. However, instead of sound, OCT employs light for tissue analysis that enables visualization of the coronary lesions with almost microscopic precision [9,10].

This tool can find high risk vulnerable plaque without angiographic or functional signs of severity, helping from misdiagnosing and under-treating these lesions, that could benefit from PCI even more than obstructive lesions without vulnerable plaque characteristics.

In an OCT substudy of the COMPLETE trial, researchers determined that half of patients had obstructive nonculprit lesions with vulnerable plaque, which could explain why complete revascularization conferred better outcomes than culprit lesion-only revascularization in the main trial. This substudy pointed out also a 20% of non-obstructive non-culprit lesions with vulnerable plaque caracteristics and up to 30% of obstructive non-culprit lesions without high risk morphology [11]. It suggest that a morphological approach to PCI in high risk patients can provide a more specific treatment compared with standard angiographic/functional approach. A correct identification of coronary plaque instability in a setting of STEMI patients could deeply impact in these patients risk of cardiovascular events, angina and re- hospitalization.

Being coronary artery disease a pandemic disease with an important impact on nations health care, a reduction in events in these patients do not impact only on patients quality of life, but on health care system resources.

Consequently, we propose a randomized controlled trial to evaluate the effective benefit of OCT guided vs complete PCI in STEMI patients with multivessels coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI and residual non culprit CAD
2. Informed consent

Exclusion Criteria:

1. Refusal or inability to provide informed consent.
2. < 18 years of age
3. Cardiogenic shock
4. Previous Coronary Artery Bypass Grafting (CABG
5. Indication for revascularization by CABG.
6. eGFR < 30 ml/min/m2
7. ULM stenosis
8. Estimated life expectancy < 3 year
9. Non culprit CTO lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 24 mounth after the recruitment in the study
  Composite endopoint of all cause mortality, cardiovascular mortality, non-fatal myocardial infarction, unplanned revascularization.

SECONDARY OUTCOMES:
Secondary efficacy end-points | 24 mounth after the recruitment in the study
  Rate of all cause mortality, cardiovascular mortality, non-fatal myocardial infarction, unplanned revascularization taking separately.

OTHER OUTCOMES:
Safety end-points | 24 mounth after the recruitment in the study
  Rate of Acute kidney injury (AKI) following OCT vs complete guided PCI, defined according to the Acute Kidney Injury Network criteria
Safety end-points | 24 mounth after the recruitment in the study
  Rate of procedural complications following each PCI: periprocedural MI defined according to the Fourth Universal Definition of Myocardial Infarction [15], arterial access site complications, AKI

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Ospedale San Luigi Gonzaga, Orbassano, Orbassano
  - Ospedale di Rivoli, Rivoli
  - AOU Città della Salute e della Scienza di Torino, Torino
  - Ospedale San Giovanni Bosco, Torino
  - Citta della Salute, Turin